CLINICAL TRIAL: NCT00966134
Title: Ghrelin, Growth Hormone and Growth Factors at High Altitude
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof Herwig Frisch, Pediatric Department
Other Study IDs: EK 411
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2009-08

CONDITIONS: Healthy; Growth Hormone
Keywords: mountain medicine; ghrelin; growth hormone; hypoxia; physiology of hormonal adaptation to high altitude
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- probands
  Interventions: Other: exposure to high altitude

INTERVENTIONS:
Other: exposure to high altitude

SUMMARY:
Regulation of ghrelin, growth hormone and growth factors at high altitude and their change during ascent to high altitude has not been studied in depth yet. The study includes 33 volunteers (12f) investigated at sea level, 4 days after ascent to 3440m and 14 days after ascent to 5400-5900m.

The investigators hypothesized that during ascent growth hormone levels would increase to compensate for the higher energy needs at high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and good physical fitness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Caucasians from an Alpinist association
Sampling Method: Non-Probability Sample
Dates: Start 2002-04; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Ghrelin, growth hormone, insulin-like growth factor I (IGF-I), IGF binding protein 1 (IGFBP1), IGF binding protein 2 (IGFBP2), IGF binding protein 3 (IGFBP3), acid-labile subunit (ALS), insulin, prolactin | 14 days